CLINICAL TRIAL: NCT04900987
Title: Application of Steri-strips for Reducing the Duration of Post Procedure Radial Artery Compression Via Conventional Pneumatic Transradial Band: An Open-label Randomized Controlled Trial
Brief Title: Steri-strips for Reducing Radial Artery Compression Duration
Acronym: RACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Kamran Ahmed Khan, Assistant Professor of Cardiology, National Institute of Cardiovascular Diseases, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ERC-29/2021
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Radial artery; TR Band; Steri-strips; Coronary angiogram; Radial patency
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: patients will be randomly assigned in a 1:1 manner to radial arterial compression with conventional pneumatic TR band alone and radial arterial compression with pneumatic TR band mechanical compression with use of clean sterile steri-strips.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment group (Experimental): After putting adequate manual pressure proximal to radial puncture site, dry and sterile application of steri-strip followed by pneumatic TR band for 1 to 2 hour.
  Interventions: Device: Steri-strips
- Control group (No Intervention): Application of pneumatic TR band alone for 4 hours as per usual practice

INTERVENTIONS:
Device: Steri-strips — Pneumatic TR band compression with use of steri-strips
  Arms: Treatment group

SUMMARY:
The duration of radial artery compression with the use of steri-strips may become much shorter than the duration of using the conventional pneumatic TR band alone for achieving hemostasis. Consequently, the frequency of radial artery occlusion (RAO) will be much lower and post procedure patency of radial artery will be higher along with significant alleviation of pain duration.

Steri-strips is a kind of sterile adhesive tape used to approximate the clean and superficial wound or surgical incision as an alternate of stitch. Its ability to keep the radial puncture site incision approximated will lead to lesser chances of platelet plug disruption or displacement at the entry site and will hasten the process of hemostasis. The use of steri-strips unlikely to have adverse consequences as it is going to be used as an assist to the usual conventional method. In a study conducted by Faravash et al. in 2016, showed significant reduction in the area of post-rhinoplasty ecchymosis in lower lid, malar and cheek soft tissues with use of steri-strips with no reported safety concerns.

Therefore, the aim of this study is to compare duration of radial artery compression by conventional method using the pneumatic TR band alone and with use of surgical steri-strips for achieving hemostasis with patency of radial artery after transradial coronary angiography along with reduction of pain duration due to arterial compression.

DETAILED DESCRIPTION:
Study population: patients undergoing coronary angiography through transradial approach. Study groups: patients will be randomly assigned in a 1:1 manner to radial arterial compression with conventional pneumatic TR band alone and radial arterial compression with pneumatic TR band mechanical compression with use of clean sterile steri-strips.

Treatment group. Pneumatic TR band compression with use of steri-strips

Control group. Pneumatic TR band compression alone

Method of radial artery compression after sheath removal:

Conventional mechanical compression: Application of pneumatic TR band alone for 4 hours.

Mechanical compression with use of steri-strips: After putting adequate manual pressure proximal to radial puncture site, dry and sterile application of steri-strip followed by pneumatic TR band for 1 hour.

END POINTS:

Primary endpoint will be the time duration of achieving hemostasis with radial artery patency

Secondary endpoint will be Hematoma or Bleeding

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary angiography through transradial approach
* Either gender with age ≥18 years
* Positive Barbeau test (type A to C)

Exclusion Criteria:

* Patients refuse to give consent
* Negative Barbeau test (type D)
* Patients with bleeding diathesis or on oral anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mean of | Immediately after removal of TR band
  Time duration of achieving hemostasis
Number of Participants with | After 24 hour of removal of TR band
  Radial artery patency

SECONDARY OUTCOMES:
Number of Participants with | Immediately after removal of TR band
  Hematoma
Number of Participants with | Immediately after removal of TR band
  Bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Farahvash MR, Khorasani G, Mahdiani Y, Taheri AR. The Effect of Steri-Strip Dressing on Patients' Satisfaction and Reduction of Ecchymosis in Lower Eyelid, Malar and Cheek Following Rhinoplasty. World J Plast Surg. 2016 Jan;5(1):51-7. PMID 27308241